CLINICAL TRIAL: NCT02060877
Title: How Burdensome is the Diagnostic Phase ? Distress and Quality of Life in Patients Suspected of Having a (Serious) Lung Disease
Brief Title: Distress and Quality of Life During the Diagnostic Phase of a Suspected Serious Lung Disease
Acronym: DIADISS
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: End-of-Life Research Group (Other)
Responsible Party: Principal Investigator, Kathleen Belien, Study Coordinator Thoracale Oncologie Groep Antwerpen, Universiteit Antwerpen
Other Study IDs: TOGA-2013; B300201419606 (Registry Identifier: Belgisch registratienummer)
Record Dates: First submitted 2014-02-04; First posted 2014-02-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Suspected Lung Cancer
Keywords: suspected lung cancer; diagnostic work-up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients suspected of having lung cancer: observational study, there is no study intervention, only patient questionnaires
  Interventions: Other: observational study: use of patient questionnaires

INTERVENTIONS:
Other: observational study: use of patient questionnaires — observational study, there is no study intervention, only patient questionnaires

SUMMARY:
The purpose of this study is to gain insight in the distress experience and quality of life of patients suspected of having a serious lung disease during the diagnostic phase and the period between diagnosis and start of treatment

DETAILED DESCRIPTION:
A life-threatening disease often leads to distress, an emotional experience that can interfere with coping. Studies in lung cancer patients show high prevalence of distress during the course of the disease. However until now, very few research was done during the diagnostic workup. This prospective study will describe and explore distress, quality of life and illness perception in lung cancer patients during the diagnostic period until first follow-up visit 4 weeks after start of therapy. Patient reported questionnaires will be used.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory patient
* imaging suggestive of lung cancer
* written informed consent
* able to complete questionnaires

Exclusion Criteria:

* solitary pulmonary nodule
* previous diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with abnormal imaging suggestive of lung cancer consulting a pulmonologist
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
longitudinal assessment of distress | at time of suspected lung cancer, at time of diagnosis, at time of treatment start, 4 weeks after treatment start
  patient reported questionnaire (distress barometer)
longitudinal assessment of quality of life | at time of suspected lung cancer, at time of diagnosis, at time of treatment start, 4 weeks after treatment start
  patient reported questionnaire (EORTC QLQ-C30 + lung cancer module)
longitudinal assessment of illness perception | at time of suspected lung cancer, at time of diagnosis, at time of treatment start, 4 weeks after treatment start
  patient reported questionnaire (Brief-Illness Perception questionnaire)
duration of diagnostic phase and period between diagnosis and treatment start | date of suspected lung cancer, date communication of diagnosis, date of treatment start

SECONDARY OUTCOMES:
explore which factors are associated with distress, quality of life and illness perception | first visit suspected lung cancer, communication of diagnosis, treatment start, 4 weeks after treatment start
  potential associated factors include patient demographic characteristics, performed diagnostic procedures, disease and treatment characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Paul Van Royen, Principal Investigator — Universiteit Antwerpen
Locations (8):
- Belgium (8):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - AZ Monica, Antwerp
  - Gasthuis Zusters Antwerpen, Antwerp
  - Universiteit Antwerpen, Antwerp
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - AZ St Jozef, Bornem
  - AZ Maria Middelares Sint Jozef, Ghent
  - AZ Herentals, Herentals

IPD SHARING:
Plan to Share IPD: No